CLINICAL TRIAL: NCT04078230
Title: Regional or Extend LymphAdenectomy During Resection of Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHCC-china
Record Dates: First submitted 2019-08-26; First posted 2019-09-06 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: resectable intrahepatic cholangiocarcinoma
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extend LymphAdenectomy (Experimental): Expanded lymph node dissection for right liver tumors included stations 12, 8, and 13, and stations 12, 1, 3, 7, and 8 for left liver tumors
  Interventions: Procedure: Extend LymphAdenectomy
- Regional LymphAdenectomy (No Intervention): Regional lymph node dissection for intrahepatic cholangiocarcinoma included station 12.

INTERVENTIONS:
Procedure: Extend LymphAdenectomy — Expanded lymph node dissection for right liver tumors included stations 12, 8, and 13, and stations 12, 1, 3, 7, and 8 for left liver tumors
  Arms: Extend LymphAdenectomy

SUMMARY:
Intrahepatic cholangiocarcinoma (ICC) is one of the common malignant tumors. Lymph node metastasis is an important factor affecting the poor prognosis of intrahepatic cholangiocarcinoma. The eighth edition of the AJCC guidelines recommends at least 6 lymph nodes to be used for staging. The American Hepatobiliary and Pancreatic Association also recommends the removal of hilar lymph nodes as part of the radical surgery for intrahepatic cholangiocarcinoma. However, some scholars have found that patients with regional lymph nodes have similar survival rates. This contradictory result has prompted more scholars to conduct clinical research to explore the necessity and standardization of lymph node dissection in intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Expanding lymph node dissection can theoretically obtain more lymph node dissection. Obtaining enough lymph nodes can improve the accuracy of AJCC staging and accurately determine prognosis. However, it is unclear whether it will improve the prognosis of patients with lymph node dissection. According to literature reports and related studies, expanded lymph node dissection for right liver tumors included stations 12, 8, and 13, and left lymphoma expanded lymph node dissection includedstations 12, 1, 3, 7, and 8.

In summary, standardize the extent of lymph node dissection in intrahepatic cholangiocarcinoma, and obtain enough lymph node dissection under the premise of controlling the complication rate, which is helpful for accurate TNM staging, accurate judgment of prognosis and improvement of survival time. Improve prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age and ≤80 years of age;
* Preoperative imaging and laboratory examination for intrahepatic cholangiocarcinoma, intraoperative frozen and postoperative pathology confirmed as intrahepatic cholangiocarcinoma; preoperative imaging assessment is resectable;
* No obvious lymph node metastasis in preoperative imaging; or negative intraoperative lymph node biopsy
* Liver function Child-Turcotte-Pugh score A-B grade;
* Residual liver volume >30%; can tolerate radical hepatectomy
* The patient has autonomy, understands and voluntarily signs the written informed consent and is able to complete the follow-up plan;
* Sign the written informed consent form prior to the test screening.

Exclusion Criteria:

* The patient has obvious heart, lung, brain and kidney dysfunction that affects the treatment of intrahepatic cholangiocarcinoma;
* The patient has a history of other malignant tumors;
* Liver function Child-Turcotte-Pugh score C;
* The investigator determined that it was not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 5 years after surgery
  disease free survival

SECONDARY OUTCOMES:
3-year Overall survival (OS) | 3 years after surgery
  3-year overall survival
Rate of Postoperative Complications (PC) | From the date of surgery to stitches off (up to 2 month)
  Postoperative Complications
5-year Overall survival (OS) | 5 years after surgery
  5-year Overall survival

CONTACTS AND LOCATIONS:
Locations (13):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States
- China (12):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Renji Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Zhong Shan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hanzhou, Zhejiang
  - Zhejiang cancer hospital, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Njei B. Changing pattern of epidemiology in intrahepatic cholangiocarcinoma. Hepatology. 2014 Sep;60(3):1107-8. doi: 10.1002/hep.26958. Epub 2014 Jul 28. No abstract available. PMID 24327308
- [Result] Zhang XF, Chakedis J, Bagante F, Chen Q, Beal EW, Lv Y, Weiss M, Popescu I, Marques HP, Aldrighetti L, Maithel SK, Pulitano C, Bauer TW, Shen F, Poultsides GA, Soubrane O, Martel G, Groot Koerkamp B, Guglielmi A, Itaru E, Pawlik TM. Trends in use of lymphadenectomy in surgery with curative intent for intrahepatic cholangiocarcinoma. Br J Surg. 2018 Jun;105(7):857-866. doi: 10.1002/bjs.10827. Epub 2018 Apr 14. PMID 29656380
- [Result] Weber SM, Ribero D, O'Reilly EM, Kokudo N, Miyazaki M, Pawlik TM. Intrahepatic cholangiocarcinoma: expert consensus statement. HPB (Oxford). 2015 Aug;17(8):669-80. doi: 10.1111/hpb.12441. PMID 26172134
- [Result] Kim DH, Choi DW, Choi SH, Heo JS, Kow AW. Is there a role for systematic hepatic pedicle lymphadenectomy in intrahepatic cholangiocarcinoma? A review of 17 years of experience in a tertiary institution. Surgery. 2015 Apr;157(4):666-75. doi: 10.1016/j.surg.2014.11.006. Epub 2015 Feb 12. PMID 25682172
- [Result] Shimada M, Yamashita Y, Aishima S, Shirabe K, Takenaka K, Sugimachi K. Value of lymph node dissection during resection of intrahepatic cholangiocarcinoma. Br J Surg. 2001 Nov;88(11):1463-6. doi: 10.1046/j.0007-1323.2001.01879.x. PMID 11683741
- [Result] Lendoire JC, Gil L, Imventarza O. Intrahepatic cholangiocarcinoma surgery: the impact of lymphadenectomy. Chin Clin Oncol. 2018 Oct;7(5):53. doi: 10.21037/cco.2018.07.02. Epub 2018 Jul 17. PMID 30180752
- [Result] Ribero D, Pinna AD, Guglielmi A, Ponti A, Nuzzo G, Giulini SM, Aldrighetti L, Calise F, Gerunda GE, Tomatis M, Amisano M, Berloco P, Torzilli G, Capussotti L; Italian Intrahepatic Cholangiocarcinoma Study Group. Surgical Approach for Long-term Survival of Patients With Intrahepatic Cholangiocarcinoma: A Multi-institutional Analysis of 434 Patients. Arch Surg. 2012 Dec;147(12):1107-13. doi: 10.1001/archsurg.2012.1962. PMID 22910846
- [Result] Doussot A, Lim C, Gomez-Gavara C, Fuks D, Farges O, Regimbeau JM, Azoulay D; AFC-IHCC Study Group. Multicentre study of the impact of morbidity on long-term survival following hepatectomy for intrahepatic cholangiocarcinoma. Br J Surg. 2016 Dec;103(13):1887-1894. doi: 10.1002/bjs.10296. Epub 2016 Sep 15. PMID 27629502